CLINICAL TRIAL: NCT05901350
Title: The Correlation of Reduction of Levodopa and Non-motor Symptoms of Parkinson's Disease After Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Levodopa reduction after DBS
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease; Visual Impairment
Keywords: Deep Brain Stimulation; Levodopa
MeSH Terms: conditions — Parkinson Disease; Vision Disorders | interventions — Levodopa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levodopa Reduction Group After STN-DBS (No Intervention): Patients in this group started to reduce levodopa dose 1 months after STN-DBS
- Levodopa non-Reduction Group After SNT-DBS (Experimental): Patients in this group did not reduce levodopa dose until 12 months after STN-DBS
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa — Some patients did not reduced the dose of levodopa after STN-DBS comparing to some without reducing the dose.
  Arms: Levodopa non-Reduction Group After SNT-DBS

SUMMARY:
Patients with parkinson disease (PD) usually reduced the dose the levodopa after received deep brain stimulation (DBS). However, studies seldomly mentioned about the influences on non-motors systems after the reduction. Our study focused on the changes after DBS and attribute them to the levodopa variety.

DETAILED DESCRIPTION:
We calculated that group sample sizes of 126 patients (63 in group 1; 63 in group 2) would provide 80% power to reject the null hypothesis of equal means when the mean difference is -5(10-15) with standard deviations of 10 for test group and 10 for control group at a two-sided alpha of 0.05. Given an anticipated dropout rate of 20%, total sample size required is 158 (79 in reduction; 79 in non-reduction group).

Written informed consent was obtained from all participants. After the baseline measurement, we informed the eligible patients the assigned randomization group with sealed opaque envelopes marked with the inpatient numbers .

Within 12 months after STN-DBS, the LEDD of the intervention group was consistent with that before operation, and gradually decreased under the guidance of physician according to the expert consensus of DBS after 12 months. The compliance problem was solved by determining the actual number of antiparkinsonian medications returned by participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants underwent neuro-ophthalmologic examinations, including ocular fundus photography, automated perimetry, and OCT. Patients undergoing deep brain stimulation (DBS) took an extra VIPD-Q after the operation.

Exclusion Criteria:

* secondary causes of parkinsonism, prior brain surgery (except DBS), glaucoma, intraocular surgery, diabetes and other diseases affecting the visual field or neurologic systems, and the current use of medications affecting visual function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
VIPD-Q scores after STN-DBS | 12 months after STN-DBS
  The VIPD-Q scores was recorded 12 months after STN-DBS

SECONDARY OUTCOMES:
RNFL thickness | 12 months after STN-DBS
Vessel density in ocular fundus | 12 months after STN-DBS
Saccades with DBS on status | 1 months after STN-DBS

CONTACTS AND LOCATIONS:
Overall Officials: chao zhang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Chao Zhang, Jinan, Shandong, China